CLINICAL TRIAL: NCT04634526
Title: Prospective Clinical Study of Intraoperative Assessment of Resection Margin of Colo-Rectal Cancer Liver Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oncology Institute of Vojvodina (Other Government)
Responsible Party: Principal Investigator, Mladjan Protic, Head of Department of Surgery, Oncology Institute of Vojvodina
Other Study IDs: No 4/18/1-972-9
Record Dates: First submitted 2020-11-10; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Liver Metastasis Colon Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective single arm double-blind study approved by the Ethics Committee of the institution, will be conducted on at the Oncology Institute of Vojvodina in Sremska Kamenica, Serbia. Patients with colo-rectal cancer liver metastases (CRLM) is presented to the multi-disciplinary team (MDT).Screening and enrolment is conducted after established of indication for resection. The surgeons assesses resection margin (RM) for every resected liver specimen (RLS) intra-operatively by inspection and palpation. These data will be compared with pathological RM examination as a "gold standard". Resection margin of 1 mm or more will be rated as negative RM (RM-) otherwise RM is positive (RM+). Taking the result of the pathohistological examination as "gold standard" it is determined that RM is true positive when the pathologist and surgeon agreed that the RM is positive. False negative RM is when the surgeon assesses RM as negative and pathologist as positive. The sensitivity of the surgical assessment of RM+ is defined as the rate of RM+ which was correctly identified. True negative RM is determined when the pathologist and surgeon agreed that it is negative RM. False positive RM defined when the surgeon assessed RM as positive, but pathologist found that it was RM-. The specificity of the surgical assessment of RM is defined as the rate of RM- which is correctly identified. Total accuracy represents the rate of correctly recognized positive and negative RM, relative to the total number of samples. Agreement between surgeon and pathologists finding will be analyzed as well as difference between them. Disease recurrence and disease-free survival (DFS) will be analyzed by RM.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Preoperative diagnosis of liver metastases of colorectal adenocarcinoma
* Indication for surgical resection of liver metastases of colorectal adenocarcinoma

Exclusion Criteria:

* RM is not defined by surgeons and pathologists as positive or negative
* Surgical resections and application of ablative procedures at the same time
* Surgery for relapse of CRLM, if the first CRLM surgery is performed before this study start
* Resection was not done from any reason

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with liver resection for liver metastases or colo-rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of R1 cases assessed by surgeon | at the operation
  Resection margin defined by surgeon could be negative (R0), positive without residual tumor (R1) and positive with residual tumor (R2)

SECONDARY OUTCOMES:
Recurrence rate | up to 5-years
  Percentage of patients with recurrence of disease
Disease free survival | up to 5-years
  Time period from operation to the disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mladjan Protic, Principal Investigator — Oncology Institute of Vojvodina
Locations (1):
- Oncology Institute of Vojvodina, Kamenitz, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Protic M, Krsmanovic O, Solajic N, Kukic B, Nikolic I, Bogdanovic B, Radovanovic Z, Kresoja M, Mannion C, Man YG, Stojadinovic A. Prospective Non-Randomized Study of Intraoperative Assessment of Surgical Resection Margin of Colo-Rectal Liver Metastases. J Cancer. 2021 Apr 30;12(12):3701-3714. doi: 10.7150/jca.58580. eCollection 2021. PMID 33995645